CLINICAL TRIAL: NCT01366976
Title: Inhibition of Lipid Peroxidation During Cardiopulmonary Bypass
Brief Title: Inhibition of Lipid Peroxidation During Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Mias Pretorius, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110423
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Cardiopulmonary Bypass Induced Lipid Peroxidation
Keywords: oxidative stress; cardiopulmonary bypass; acetaminophen; hemolysis
MeSH Terms: conditions — Hemolysis | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Acetaminophen
- Acetaminophen (Active Comparator): Acetaminophen will ge given as 1g every 6 hours for 4 doses over a 24 hours study period
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 1g every 6 hours for 4 doses over 24 hours
  Other Names: Tylenol

SUMMARY:
Acute kidney injury is a major complication of cardiac surgery requiring cardiopulmonary bypass (CPB). Hemolysis and rhabdomyolysis frequently occur during CPB. Hemolysis leads to an increase in free hemoglobin, whereas rhabdomyolysis leads to an increase in myoglobin. Free plasma hemoglobin and myoglobin have been shown to be independent predictors of the acute kidney injury that results from CPB. When these hemeproteins are released into the plasma, they undergo redox cycling, generating radical species that initiate lipid peroxidation and a cascade of oxidative damage to cellular membranes, notably in the kidney. F2-isoprostanes and isofurans are sensitive and specific markers of oxidative stress in vivo, and are increased after CPB, particularly in those patients with acute kidney injury. Acetaminophen inhibits the lipid peroxidation catalyzed by myoglobin and hemoglobin. Moreover, in an animal model of rhabdomyolysis-induced kidney injury, acetaminophen significantly attenuated the decrease in creatinine clearance compared to control. The current proposal tests the central hypothesis that acetaminophen will attenuate the lipid peroxidation associated with the hemolysis and rhabdomyolysis that occur in patients undergoing CPB. Demonstration that acetaminophen inhibits the lipid peroxidation resulting from CPB would provide a rationale for a prospective randomized trial to test the hypothesis that acetaminophen will reduce the acute kidney injury that results from CPB.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, 18 to 80 years of age, scheduled for elective cardiac surgery requiring CPB
2. For female subjects, the following conditions must be met:

postmenopausal for at least 1 year, or status-post surgical sterilization, or if of childbearing potential, utilizing adequate birth control and a negative urine beta-hcg prior to drug treatment

Exclusion Criteria:

1. Allergic reaction to ApAP (acetaminophen)
2. Evidence of severe hepatic impairment (history of liver cirrhosis or total bilirubin >2.0mg/dl)
3. Impaired renal function (serum creatinine >2.0 mg/dl)
4. Emergency surgery
5. Pregnancy
6. Breast-feeding
7. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
8. History of alcohol or drug abuse
9. Treatment with any investigational drug in the 1 month preceding the study
10. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
11. Inability to comply with the protocol, e.g. uncooperative attitude and unlikelihood of completing the study
12. History or evidence of active asthma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mias Pretorius, MBChB, MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Billings FT 4th, Ball SK, Roberts LJ 2nd, Pretorius M. Postoperative acute kidney injury is associated with hemoglobinemia and an enhanced oxidative stress response. Free Radic Biol Med. 2011 Jun 1;50(11):1480-7. doi: 10.1016/j.freeradbiomed.2011.02.011. Epub 2011 Feb 18. PMID 21334433
- [Background] Boutaud O, Moore KP, Reeder BJ, Harry D, Howie AJ, Wang S, Carney CK, Masterson TS, Amin T, Wright DW, Wilson MT, Oates JA, Roberts LJ 2nd. Acetaminophen inhibits hemoprotein-catalyzed lipid peroxidation and attenuates rhabdomyolysis-induced renal failure. Proc Natl Acad Sci U S A. 2010 Feb 9;107(6):2699-704. doi: 10.1073/pnas.0910174107. Epub 2010 Feb 1. PMID 20133658
- [Derived] Billings FT 4th, Petracek MR, Roberts LJ 2nd, Pretorius M. Perioperative intravenous acetaminophen attenuates lipid peroxidation in adults undergoing cardiopulmonary bypass: a randomized clinical trial. PLoS One. 2015 Feb 23;10(2):e0117625. doi: 10.1371/journal.pone.0117625. eCollection 2015. PMID 25705899

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled by the research nurse at the time of the preoperative evaluation for surgery. The study period was from January 2012 until April 2013.
Pre-assignment Details: Patients were excluded for the following reasons: 1) allergy to acetaminophen, 2) evidence of severe hepatic impairment (history of liver cirrhosis or total bilirubin >2.0mg/dL) 3) evidence of impaired renal function (serum creatinine >2.0mg/dL) or 4) pregnancy.
Groups:
- Acetaminophen: IV acetaminophen 1g every 6 hours for 4 doses over a 24 hours study period
- Placebo: Saline in equivalent volume as study drug
Period: Overall Study
Arm/Group | Acetaminophen | Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients were eligible for the study if he/she was 18-80 years of age and undergoing elective cardiac surgery requiring cardiopulmonary bypass.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.5 [49 to 68.4] | 61.0 [54 to 67.8] | 63 [51.75 to 67.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 20 | 16 | 36
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Plasma Isofuran Concentrations
Description: Plasma isofuran concentrations as a measure of lipid peroxidation
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: pg/mL
Groups:
- Placebo: Saline infusion
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 30 | 30
pg/mL
  baseline | 61.5 (6.8) | 67.7 (5.97)
  30min of bypass | 72.1 (7.37) | 82.7 (6.02)
  60min of bypass | 83.4 (7.55) | 110.8 (13.21)
  post-bypass | 82.9 (9.71) | 96.1 (8.22)
  ICU | 85.3 (8.53) | 88.0 (8.81)
  postoperative day 1 | 70.4 (8.45) | 68.5 (6.21)
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; We hypothesized that acetaminophen would reduce peak isofuran concentrations by 22 pg/mL (40% reduction from peak concentrations). If the true difference in the acetaminophen and placebo group means is 22 pg/mL (SD=30 pg/mL), we would need to study 30 experimental subjects and 30 control subjects to be able to reject the null hypothesis that the population means of the acetaminophen and placebo groups are equal with probability (power) 0.8; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis

2. Secondary Outcome: Urinary NGAL (Neutrophil Gelatinase-associated Lipocalin)
Description: Changes in urinary NGAL (neutrophil gelatinase-associated lipocalin) as marker of acute kidney injury
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 30 | 30
ng/mL
  baseline | 19.21 (6.7) | 23.2 (8.4)
  pos-bypass | 145.8 (49.6) | 138.4 (43.5)
  postoperative day 1 | 46.04 (25.5) | 16.8 (2.4)

3. Primary Outcome: Plasma F2-isoprostane Concentrations
Description: Plasma F2-isoprostane concentrations as a measure of lipid peroxidation
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 30 | 30
pg/mL
  baseline | 27.8 (3.3) | 30.6 (3.5)
  30min of bypass | 45.8 (3.7) | 49.1 (4.9)
  60min of bypass | 52.0 (5.3) | 52.8 (6.0)
  post-bypass | 34 (2.9) | 48.4 (10.2)
  ICU | 32.0 (3.1) | 47.5 (9.9)
  postoperative day 1 | 26.5 (2.9) | 26.0 (2.6)
Statistical Analysis 1: Comparison: Acetaminophen vs Placebo; Test type: Superiority or Other; p = 0.12, Mixed Models Analysis

4. Secondary Outcome: Serum Creatinine
Description: Serum creatinine measured over a 72 hour period
Time Frame: 72 hours
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Acetaminophen | Placebo
Number analyzed (Participants) | 30 | 30
mg/dL
  baseline | 0.98 (0.04) | 0.94 (0.03)
  postoperative day 1 | 0.89 (0.04) | 0.90 (0.04)
  postoperative day 2 | 0.96 (0.04) | 0.96 (0.04)
  postoperative day 3 | 0.93 (0.04) | 0.88 (0.05)

ADVERSE EVENTS:
Time Frame: Duration of hospitalization up to 2 weeks
Arm/Group | Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/30 | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen (N=30) | Placebo (N=30)
Postoperative atrial fibrillation (Cardiac disorders) | 4 (4) | 4 (4)
Re-exploration for bleeding (Surgical and medical procedures) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
The exploratory analysis of acute kidney injury (AKI) was limited by the low incidence of postoperative AKI in the current study, so we were underpowered to detect small differences in creatinine or NGAL concentrations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No